CLINICAL TRIAL: NCT01131221
Title: Vitamin D Insufficiency and Follicular Lymphoma Prognosis
Brief Title: S8947-9800-9911-0016A Vitamin D Insufficiency in Determining Prognosis in Patients With Newly Diagnosed Follicular Lymphoma
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000671527; SWOG-S8947-9800-9911-0016-A
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of serum from patients with cancer in the laboratory may help doctors identify and learn more biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying vitamin D insufficiency in determining prognosis in patients with newly diagnosed follicular lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the role of pre-treatment serum 25(OH)D with regard to progression-free survival and objective response among patients with newly diagnosed follicular lymphoma, within the context of a uniformly treated and evaluated Phase III clinical trial in the modern therapeutic era.

OUTLINE: This is a multicenter study.

Pre-treatment serum samples are analyzed for 25(OH)D levels to determine vitamin D sufficiency or insufficiency.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed CD20+ follicular lymphoma
* Enrolled on clinical trial SWOG-S0016, SWOG-9800, or SWOG-9911
* Pre-treatment serum available through SWOG-8947

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients enrolled in S8947-9800-9911-0016 consenting to banking
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | retrospective

SECONDARY OUTCOMES:
Objective response (confirmed and unconfirmed complete and partial responses) | retrospective

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Friedberg, MD, Principal Investigator — James P. Wilmot Cancer Center